CLINICAL TRIAL: NCT07391241
Title: A Randomised, Double-blind, Placebo-controlled, 4-way Cross-over Trial Studying the Efficacy and Safety of Single Dose Administration of Pudafensine in Vulvodynia (Provoked Vestibulodynia).
Brief Title: A Phase 2 Study to Evaluate the Efficacy and Safety of Pudafensine in Vulvodynia (Provoked Vestibulodynia)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Initiator Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IP2015CS05
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose_1 (Experimental): Pudafensine
  Interventions: Drug: Pudafensine
- Dose_2 (Experimental): Pudafensine
  Interventions: Drug: Pudafensine
- Dose_3 (Experimental): Pudafensine
  Interventions: Drug: Pudafensine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Pudafensine

INTERVENTIONS:
Drug: Pudafensine — Pudafensine

SUMMARY:
The study (IP2015CS05) is a randomised, double-blind, placebo-controlled, 4-way cross-over trial studying the efficacy and safety of single dose administration of pudafensine in vulvodynia (provoked vestibulodynia) patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant with vulvodynia (provoked vestibulodynia).

Exclusion Criteria:

* Women with vulvar pain caused by a specific disorder:

  1. Infectious (e.g. recurrent candidiasis, herpes).
  2. Inflammatory (e.g. lichen sclerosus, lichen planus, immunobullous disorders).
  3. Neoplastic (e.g. Paget disease, squamous cell carcinoma).
  4. Neurologic (e.g. postherpetic neuralgia, nerve compression or injury, neuroma).
  5. Trauma (e.g. female genital cutting, obstetrical).
  6. Iatrogenic (e.g. postoperative, chemotherapy, radiation).
  7. Hormonal deficiencies (e.g. genitourinary syndrome of menopause (vulvovaginal atrophy), lactational amenorrhea).
* History or current diagnosis of significant pelvic floor dysfunction.
* Co-morbid pelvic pain conditions including pain due to pelvic fractures, pelvic girdle pain or post-partum pelvic pain (to avoid confounding pain outcomes).
* History or current diagnosis of pelvic inflammatory disease.
* History or current diagnosis of endometriosis.
* History or current diagnosis of interstitial cystitis.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the effect of pudafensine on pain in the vaginal vestibule (vestibular pain threshold) using the Vestibular Pain Threshold Test | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Abimbola Babajide, Dr, Principal Investigator — MAC, UK
Locations (1):
- MAC, Blackpool, United Kingdom